CLINICAL TRIAL: NCT00997633
Title: Single-photon Emission Computed Tomography for Prediction of Treatment Results in Sequential Intraperitoneal Chemotherapy at Peritoneal Carcinomatosis
Brief Title: Single-photon Emission Computed Tomography (SPECT) to Predict Peritoneal Chemotherapy
Status: Completed | Type: Observational
Sponsor: Uppsala University (Other)
Responsible Party: Haile Mahteme, MD PhD, Dept of Surgical Sciences, Section of Surgery, Uppsala University, Sweden
Other Study IDs: SPECT IK1991:5
Record Dates: First submitted 2009-10-16; First posted 2009-10-19 (Estimated); Last update posted 2009-10-19 (Estimated); Status verified 2009-10

CONDITIONS: Peritoneal Carcinomatosis
Keywords: Intraperitoneal volume; peritoneal carcinomatosis; cytoreductive surgery; SPECT; intraperitoneal chemotherapy
MeSH Terms: conditions — Peritoneal Neoplasms

STUDY DESIGN:
Observational Model: Case-Only
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Peritoneal carcinomatosis: Patients undergoing cytoreductive surgery and intraperitoneal chemotherapy treatment

SUMMARY:
SPECT was performed in 51 patients after cytoreductive surgery in combination with intraperitoneal chemotherapy. The detected volume was compared to the number of subsequent sequential postoperative intraperitoneal chemotherapy courses that could be performed without further surgical intervention. SPECT data was found to predict feasibility of sequential postoperative intraperitoneal chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Cytoreductive surgery and intraperitoneal chemotherapy
* Single-Photon Emission Computed Tomography (SPECT) before the second course of treatment

Ages: 14 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who had undergone cytoreductive surgery and intraperitoneal chemotherapy (SPIC) at the Dept of Surgical Sciences, Uppsala University Hospital in the time period between May 1991 and August 2004.
Sampling Method: Non-Probability Sample
Enrollment: 51 (Actual)
Dates: Start 1991-05; Primary Completion 2004-08 (Actual); Study Completion 2004-08 (Actual)

PRIMARY OUTCOMES:
Detected volume measured by SPECT compared to the number of subsequent sequential postoperative intraperitoneal chemotherapy courses

SECONDARY OUTCOMES:
The relationship between SPECT, feasibility of SPIC (intraperitoneal chemotherapy), and clinical variables

CONTACTS AND LOCATIONS:
Overall Officials: Haile Mahteme, MD PhD, Principal Investigator — Dept of Surgical Sciences, University Hospital, Uppsala, Sweden
Locations (1):
- Dept of Surgical Sciences, Section of Surgery, S-751 85 Uppsala, Sweden